CLINICAL TRIAL: NCT05847842
Title: Comparison of the Effects of Local Anesthetic Infiltration and Different Fascial Plane Blocks on Postoperative Recovery Quality and Pain in Inguinal Hernia Repair
Brief Title: Comparison of Local Anesthetic Infiltration and Different Fascial Plane Blocks in Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Gulay ERDOGAN KAYHAN, Professor Doctor, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESOGUhernia
Record Dates: First submitted 2023-04-18; First posted 2023-05-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain; Inguinal Hernia; Local Infiltration; Quality of Recovery; Quadratus Lumborum Block; Transversus Abdominis Plane Block
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Q (Active Comparator): Anterior quadratus lumborum block
  Interventions: Procedure: Anterior quadratus lumborum block
- Group T (Active Comparator): Transversus abdominis plane block
  Interventions: Procedure: Transversus abdominis plane block
- Group L (Active Comparator): Local infiltration
  Interventions: Procedure: Local infiltration

INTERVENTIONS:
Procedure: Anterior quadratus lumborum block — 20 mL of 0.25% bupivacaine will be given
  Arms: Group Q
Procedure: Transversus abdominis plane block — 20 mL of 0.25% bupivacaine will be given
  Arms: Group T
Procedure: Local infiltration — 20 mL of 0.25% bupivacaine will be given
  Arms: Group L

SUMMARY:
In this study, quadratus lumborum block (QLB), transversus abdominis plane (TAP) block, and local anesthetic infiltration will be performed preoperatively in patients who will undergo unilateral inguinal herniorrhaphy operation under general anesthesia. Quality of recovery (QoR-15) score, postoperative acute and chronic pain levels will be evaluated.

DETAILED DESCRIPTION:
Inguinal hernia repair, one of the most common operations, causes moderate to severe postoperative pain. The postoperative pain delays patients' recovery and return to daily life, increases the rate of readmission to the hospital, and can lead to persistent postoperative pain.Procedure-specific postoperative pain management (PROSPECT) recommendations for optimal pain management have been recently updated. Accordingly, in addition to preoperative or intraoperative paracetamol and nonsteroidal anti-inflammatory analgesics, local anesthetic infiltration and/or regional analgesia techniques (ilio-inguinal nerve blocks or TAP block) with rescue opioids are recommended. Also, it has been reported that further research is needed on new regional techniques (other fascial plane blocks etc).It has been shown that QLB potentially results in extensive sensory blockade (T7-12), and in cadaver studies, the iliohypogastric and ilioinguinal nerves are constantly involved. In addition, there are studies suggesting that it provides much longer analgesia than TAP block. There are few studies on its efficacy in inguinal hernia repair that are in pediatric cases or performed in addition to central blocks. It is hypothesized that QLB may provide better and longer analgesia, may increase the quality of recovery and reduce the development of resistant chronic pain, compared to other regional methods such as local infiltration or TAP block, that proven effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo elective unilateral inguinal herniorrhaphy under general anesthesia
* American Society of Anesthesiology (ASA) physical classification I-III

Exclusion Criteria:

* Patients who will undergo laparoscopic surgery
* Previous inguinal hernia repair surgery
* A history of opioid use or pain management
* Coagulopathy or anticoagulant use
* Patients who have difficulty communicating or who are not cooperative

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Quality of recovery assessed by Quality of recovery scale (QoR-15) | Postoperative 24th hour.
  The 15-item quality of recovery (QoR-15) scale is a questionnaire used to evaluate the postoperative recovery quality of patients in the early postoperative stages. The QoR-15 score comprises 15 questions that assess 5 recovery domains, namely, physical comfort, physical independence, psychological support, emotional status, and pain. Each question is scored from 0 to 10 (0 none of the time to 10 all of the time).

SECONDARY OUTCOMES:
Postoperative pain assessed by Numerical Rating Scale (NRS) | At the 2nd, 6th, 12th, 24th and 36th hours
  Postoperative pain levels during rest and movement (from supine to sitting position) will be evaluated by Numerical rating scale (0-no pain; 10-unbearable pain)
Postoperative chronic pain assessed by Numerical Rating Scale (NRS) | Three months later the operation date
  Patients will be called by phone and the presence of chronic pain will be questioned with the Numerical Rating Scale (0-no pain; 10-unbearable pain).
Postoperative neuropathic pain assessed by Douleur neuropathic pain (DN4) scale. | Three months later the operation date
  Patients will be called by phone and the presence of neuropathic pain pain will be questioned with the Douleur neuropathic pain (DN4) scale.
  The items of the DN4 are scored based on a yes (1 point) /no (0 points) answer. This leads to a score range of 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Gulay Erdogan Kayhan, Prof Dr, Principal Investigator — Eskisehir Osmangazi University
Locations (2):
- Turkey (Türkiye) (2):
  - Eskisehir Osmangazi University Faculty of Medicine, Eskişehir
  - Eskisehir Osmangazi Universty, Eskişehir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okur O, Karaduman D, Tekgul ZT, Koroglu N, Yildirim M. Posterior quadratus lumborum versus transversus abdominis plane block for inguinal hernia repair: a prospective randomized controlled study. Braz J Anesthesiol. 2021 Sep-Oct;71(5):505-510. doi: 10.1016/j.bjane.2020.11.004. Epub 2021 Feb 10. PMID 34537121